CLINICAL TRIAL: NCT05156320
Title: Phase 3, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Apitegromab (SRK-015) in Patients With Later-Onset Spinal Muscular Atrophy Receiving Background Nusinersen or Risdiplam Therapy
Brief Title: Efficacy and Safety of Apitegromab in Patients With Later-Onset Spinal Muscular Atrophy Treated With Nusinersen or Risdiplam
Acronym: SAPPHIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scholar Rock, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRK-015-003
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Spinal Muscular Atrophy; Spinal Muscular Atrophy Type 3; Spinal Muscular Atrophy Type 2; SMA; Neuromuscular Diseases; Muscular Atrophy; Atrophy; Muscular Atrophy, Spinal; Neuromuscular Manifestations; Anti-myostatin
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophies of Childhood; Neuromuscular Diseases; Muscular Atrophy; Atrophy; Neuromuscular Manifestations | interventions — apitegromab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active treatment, randomized, double-blind, placebo-controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Main Efficacy Population (Apitegromab 10 mg/kg) (Experimental): Aged 2-12 years at Screening. Participants were randomized to receive apitegromab 10 mg/kg for up to 52 weeks.
  Interventions: Drug: Apitegromab
- Main Efficacy Population (Apitegromab 20 mg/kg) (Experimental): Aged 2-12 years at Screening. Participants were randomized to receive apitegromab 20 mg/kg for up to 52 weeks.
  Interventions: Drug: Apitegromab
- Main Efficacy Population (Placebo) (Placebo Comparator): Aged 2-12 years at Screening. Participants were randomized to receive placebo for up to 52 weeks.
  Interventions: Drug: Placebo
- Exploratory Subpopulation (Apitegromab) (Experimental): Aged 13-21 years at Screening. Participants were randomized to receive apitegromab 20 mg/kg for up to 52 weeks.
  Interventions: Drug: Apitegromab
- Exploratory Subpopulation (Placebo) (Placebo Comparator): Aged 13-21 years at Screening. Participants were randomized to receive placebo for up to 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apitegromab — Apitegromab is a fully human anti-proMyostatin monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/lambda isotype that specifically binds to human pro/latent myostatin with high affinity inhibiting myostatin activation. SRK-015 was administered every 4 weeks by intravenous (IV) infusion.
  Other Names: SRK-015
  Arms: Exploratory Subpopulation (Apitegromab); Main Efficacy Population (Apitegromab 10 mg/kg); Main Efficacy Population (Apitegromab 20 mg/kg)
Drug: Placebo — Placebo was administered every 4 weeks by intravenous (IV) infusion.
  Arms: Exploratory Subpopulation (Placebo); Main Efficacy Population (Placebo)

SUMMARY:
This Phase 3 trial (Study SRK-015-003) was conducted in patients ≥2 years old at Screening, who were previously diagnosed with later-onset spinal muscular atrophy (SMA) (i.e., Type 2 and Type 3 SMA) and were receiving an approved survival motor neuron (SMN) upregulator therapy (i.e., either nusinersen or risdiplam), to confirm the efficacy and safety of apitegromab as an adjunctive therapy to nusinersen and evaluate the efficacy and safety of apitegromab as an adjunctive therapy to risdiplam.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 2 through 21 years old at Screening.
* Documented diagnosis of 5q SMA.
* Diagnosed with later-onset SMA (i.e., Type 2 and Type 3 SMA) before receiving an approved SMN upregulator therapy (i.e., either nusinersen or risdiplam).
* Must be Nonambulatory at Screening. Nonambulatory patients must be able to sit independently (sits up straight with head erect for at least 10 seconds; does not use arms or hands to balance body or support position) per World Health Organization (WHO) motor milestones definition at Screening.
* Receiving one background therapy for SMA (i.e., either nusinersen or risdiplam) for the time period specified below and anticipated to remain on that same treatment throughout the trial:

  1. If receiving the SMN upregulator therapy nusinersen, must have completed at least 10 months of dosing (i.e., completed the loading regimen and at least 2 maintenance doses) before Screening;
  2. If receiving the SMN upregulator therapy risdiplam, must have completed at least 6 months of dosing before Screening.
* Motor Function Score (HFMSE) ≥10 and ≤45 at Screening.
* Have no physical limitations that would prevent the patient from undergoing motor function outcome measures throughout the duration of the study.
* Able to receive study drug infusions and provide blood samples through the use of a peripheral intravenous (IV) or a long-term IV access device that the patient has placed for reasons independent from the study throughout the duration of the study.
* Able to adhere to the requirements of the protocol, including travel to the study center and completing all study procedures and study visits.
* For patients who are expected to have reached reproductive maturity by the end of the study, adhere to study specific contraception requirements.

Exclusion Criteria:

* Received ZOLGENSMA® (onasemnogene abeparvovec-xioi) at any time and previous treatment with apitegromab.
* Use of invasive ventilation and tracheostomy.
* Use of chronic daytime non-invasive ventilatory support for >16 hours daily in the 2 weeks prior to dosing, or anticipated to regularly receive such daytime ventilator support chronically over the duration of the study.
* Any acute or co-morbid condition interfering with the well-being of the patient within 7 days of screening, including active systemic infection, the need for acute treatment or inpatient observation due to any reason.
* Severe scoliosis and/or contractures at screening. Based on clinical judgement, any scoliosis or contractures present must be stable over the past 6 months, anticipated to be stable for the duration of the study and not prevent the patient from being evaluated on any functional outcome measures throughout the duration of the study.
* Pregnant or breastfeeding.
* Major orthopedic or other interventional procedure, including spine or hip surgery, considered to have the potential to substantially limit the ability of the patient to be evaluated on any functional outcome measures, within 6 months prior to Screening, or anticipated for the duration of the study.
* Prior history of a hypersensitivity reaction to a monoclonal antibody (mAb) or recombinant protein bearing an Fc domain (such as a soluble receptor-Fc fusion protein), apitegromab, or excipients of apitegromab.
* Treatment with investigational drugs within 3 months prior to Screening.
* Use of therapies with potentially significant muscle effects (such as androgens, insulin-like growth factor, growth hormone, systemic beta-agonist, botulinum toxin, or muscle relaxants or muscle-enhancing supplements) or potentially significant neuromuscular effects (such as acetylcholinesterase inhibitors) within 60 days prior to screening.
* Nutritional status not stable over the past 6 months and not anticipated to be stable throughout the duration of the study.
* Patient has any other condition, which in the opinion of the Investigator may compromise safety or compliance, would preclude the patient from successful completion of the study, or interfere with the interpretation of the results.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 188 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Main Efficacy Population: Change from Baseline in Hammersmith Functional Motor Scale Expanded (HFMSE) total score. | Baseline up to 12 months.
  The HFMSE assesses the physical abilities of patients with Type 2 and Type 3 SMA. It comprises of 33 items graded on a scale of 0, 1, or 2, where 0 denotes unable, 1 denotes performed with modification or adaptation, and 2 denotes performed without modification or adaptation. The overall score is the sum of the scores for all activities with a maximum achievable score of 66. Higher scores indicate increased motor function.

SECONDARY OUTCOMES:
Main Efficacy Population: Change from Baseline in Revised Upper Limb Module (RULM) total score. | Baseline up to 12 months.
  The RULM is a 20 item assessment of upper limb function in nonambulatory patients with SMA that was performed for patients who were 30 months of age or older at baseline. The 19 scored items assess functions that relate to everyday life, such as pressing a button and picking up a token; these items are scored 0, 1, or 2, where 0 denotes unable, 1 denotes able with modification, and 2 denotes able with no modification. The maximum score achievable is 37. Higher scores increased great upper limb function.
Main Efficacy Population: Proportion of patients with ≥3-point change from Baseline in Hammersmith Functional Motor Scale Expanded (HFMSE) total score. | Baseline up to 12 months.
  The HFMSE assesses the physical abilities of patients with Type 2 and Type 3 SMA. It comprises of 33 items graded on a scale of 0, 1, or 2, where 0 denotes unable, 1 denotes performed with modification or adaptation, and 2 denotes performed without modification or adaptation. The overall score is the sum of the scores for all activities with a maximum achievable score of 66. Higher scores indicate increased motor function.
Main Efficacy Population: Change from Baseline in number of WHO motor development milestones attained at 12 months. | Baseline up to 12 months.
Main Efficacy Population and Exploratory Subpopulation combined: Incidence of Treatment Emergent Adverse Events (TEAEs) and Severe Adverse Events (SAEs) by severity. | Baseline up to 12 months.
Main Efficacy Population and Exploratory Subpopulation combined: Apitegromab concentrations in serum from blood samples. | Baseline up to 12 months.
Main Efficacy Population and Exploratory Subpopulation combined: Circulating latent myostatin concentrations in blood samples. | Baseline up to 12 months.
Main Efficacy Population and Exploratory Subpopulation combined: Presence or absence of Antidrug Antibody (ADA) against apitegromab in serum from blood samples. | Baseline up to 12 months.

CONTACTS AND LOCATIONS:
Locations (50):
- United States (26):
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Rady's Children's Hospital/UCSD, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Hospital, Orlando, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - The Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Columbia University, SMA Clinical Research Center, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
- Belgium (3):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - Chr de La Citadelle, Liège
- France (3):
  - CHU Lille - Hôpital Jeanne de Flandre, Lille
  - Hôpital Armand Trousseau, I-Motion, Paris
  - CHU Toulouse - Hopital des Enfants, Toulouse
- Germany (4):
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Essen, Essen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Dr. von Haunersches Kinderspital, Munich
- Italy (5):
  - IRCCS Istituto Giannina Gaslini, Genoa
  - A.O.U Policlinico G. Martino, Messina
  - Foundation I.R.C.C.S. Carlo Besta Neurological Institute, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Centro Clinico Nemo Pediatrico Policlinico A. Gemelli-Università Cattolica Sacro Cuore, Roma
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne w Gdańsku, Gdansk
  - Uniwersytet Medyczny im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Instytut Pomnik - Centrum Zdrowia Dziecka: CZD Warszawa, Warsaw
- Spain (2):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitario y Politécnico La Fe, Valencia
- United Kingdom (3):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - University of Oxford, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crawford TO, Servais L, Mercuri E, Kolbel H, Kuntz N, Finkel RS, Krueger J, Batley K, Young SD, Marantz JL, Song G, Yao B, Zhao G, Rossello J, Tirucherai GS, Mazzone ES, Butterfield RJ, de la Banda MGG, Seferian AM, Sansone VA, De Waele L, van der Pol WL, Cances C, Pechmann A, Darras BT; SAPPHIRE Study Group. Safety and efficacy of apitegromab in nonambulatory type 2 or type 3 spinal muscular atrophy (SAPPHIRE): a phase 3, double-blind, randomised, placebo-controlled trial. Lancet Neurol. 2025 Sep;24(9):727-739. doi: 10.1016/S1474-4422(25)00225-X. PMID 40818473